CLINICAL TRIAL: NCT06001008
Title: Validity of the Turkish Version of "Perception of Quality in Anesthesia": A Prospective Observational Cohort Study
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, dilan akyurt, Specialist of Anaesthesiology and Reanimasion Principle investigator, Samsun University
Other Study IDs: SÜKAEK-2022/5/12
Record Dates: First submitted 2023-07-29; First posted 2023-08-21 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2023-10

CONDITIONS: Patient Satisfaction
Keywords: Anesthesia; Perioperative complications; PQA
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- General or regional anesthesia: Patients who have undergone inguinal or umbilical hernia surgery
  Interventions: Other: PQA

INTERVENTIONS:
Other: PQA — PQA is a questionnaire consisting of 16 questions developed to measure the quality of anesthesia service received by patients based on their experiences. Patients will be asked to answer questions by the researcher 24 hours after surgery.

SUMMARY:
The aim of this study is to test the validity of the Perception of Quality in Anesthesia (PQA) and language compatibility.

DETAILED DESCRIPTION:
The Perception of Quality in Anesthesia (PQA) scale was developed by Hocking et al. in 2013 to measure the quality of anesthesia service received by patients who underwent surgery under anesthesia. The survey consists of 16 questions. Researchers ask patients undergoing surgery to complete the PQA questionnaire 24 hours after surgery. The researcher visits patients in hospital rooms or makes phone calls the day after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective inguinal or umbilical hernia surgery under general or regional anesthesia
* Age between 18 and 80 years
* Ability to understand the content of surveys
* Native speaker of Turkish

Exclusion Criteria:

* Emergency operation
* The need for postoperative intensive care
* Existence of mental disability
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing electiveinguinal or umbilical hernia surgery under general or regional anesthesia in Samsun University Hospital
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Construct Validity of PQA (Perception of Quality in Anesthesia) | 24 hours after the surgery
  PQA is a 16-item questionnaire that measures the satisfaction of the patient with the anesthesia approach applied in the perioperative period. Survey questions assess 5 topics: Factor A: attention/courtesy; Factor B: pain management; Factor C: knowledge/trust; Factor D: POB; and Factor E: concerns addressed. For each question, the patient is asked to answer using a five-point Likert scale. The extremes of the scale are labeled 'very poor' to 'very good' or 'definitely no' to 'definitely yes' depending on the question. Patient responses to each PQA Likert scale and visual analog questions are scored from 1 to 5. 'Absolutely no' or 'very poor' is scored as 1 and 'definitely yes' or 'very good' is scored 5.

SECONDARY OUTCOMES:
Response success rate of the PQA | 24 hours after the surgery
  Defined as success if the patient has answered all items

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa SÜREN, Study Director — Samsun University
Locations (1):
- Dilan Akyurt, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Hocking G, Weightman WM, Smith C, Gibbs NM, Sherrard K. Measuring the quality of anaesthesia from a patient's perspective: development, validation, and implementation of a short questionnaire. Br J Anaesth. 2013 Dec;111(6):979-89. doi: 10.1093/bja/aet284. Epub 2013 Aug 28. PMID 23985532